CLINICAL TRIAL: NCT06508736
Title: The Effect of Storytelling on Cyberbullying and Empathy in Adolescents
Brief Title: Cyberbullying, Empathy, and Storytelling in Adolescents
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Sultan Ayaz Alkaya, Prof., Gazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023 - 1571
Record Dates: First submitted 2024-07-06; First posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Cyberbullying
MeSH Terms: conditions — Cyberbullying

STUDY DESIGN:
Intervention Model Description: randomized trial with experimental and control groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Storytelling Grup (Experimental): Participants will receive 4 sessions of storytelling intervention with expert reviewed stories.
  Interventions: Behavioral: Storytelling
- Active Comparator Grup (Active Comparator): Participants will be trained on cyberbullying in 4 sessions.
  Interventions: Behavioral: Training

INTERVENTIONS:
Behavioral: Storytelling — It is aimed that adolescents gain behavioral change through stories.
  Arms: Storytelling Grup
Behavioral: Training — Participants will be trained on cyberbullying in 4 sessions.
  Arms: Active Comparator Grup

SUMMARY:
The type of this study is a randomized controlled experimental study. The aim of this study is to determine the effect of storytelling method on cyberbullying and empathy level in adolescents. The population of the study consisted of 5th and 6th grade middle school students. The sample of the study will consist of students involved in cyberbullying. The sample will be selected through randomization and stratified selection will be made according to gender. The students in the intervention group will receive 4 sessions of storytelling intervention. The active control group will receive 4 sessions of cyberbullying training. Questions that the research aims to answer:

Is there a difference between the intervention group and the control group in terms of cyberbullying level? Is there a difference between the intervention groups and the control group in terms of empathy level?

Participants:

The intervention group will participate in 4 sessions of storytelling intervention.

The control group will participate in 4 sessions of cyberbullying training.

ELIGIBILITY:
Inclusion Criteria:

* Family approval
* Volunteering to participate in the study.
* Being a 5th and 6th grade student
* Engaging in cyberbullying behavior

Exclusion Criteria:

* Having a diagnosis of any mental illness
* Having at least one of vision, speech and hearing disabilities
* Foreign nationality
* Being a 7th and 8th grade student
* Not engaging in cyberbullying behavior

Ages: 10 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
cyberbullying | 6 months
  It is expected that cyberbullying will decrease with storytelling. These measurements will be made with the Cyberbullying Triangle Scale. Cyberbullying Triangle Scale and Bullying, Victimization and Cyber Bystander subscales will be used in the evaluation. The assessment is done by categorizing students into various categories. These categories are: "not involved in cyberbullying, only cyber victim, only cyber bully, only cyber bystander, cyber bully and cyber victim, cyber bystander and cyber victim, cyber bystander and cyber bully, cyber bully, cyber victim and cyber bystander".

SECONDARY OUTCOMES:
empathy | 6 months
  Empathy parameter is expected to increase with storytelling. Empathy will be assessed with the Cognitive, Affective, Behavioral Empathy Scale. The Empathy Scale consists of 30 questions and three sub-factors: cognitive, affective and bodily empathy. The scale has a 3-point Likert (0 and 2) type rating. The score that can be obtained from the scale varies between 0 and 60 and the higher the score, the higher the empathy tendency.

IPD SHARING:
Plan to Share IPD: Undecided